CLINICAL TRIAL: NCT04526054
Title: Longitudinal and Comparative Study of Morphological Abnormalities of the Olfactory Bulb on MRI and Olfactometry in Anosmic Versus Normosmic COVID-19 Patients
Brief Title: Morphological Abnormalities of the Olfactory Bulb on MRI and Olfactometry in Anosmic Versus Normosmic COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: Hôpital Raymond Poincaré (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020_0057
Record Dates: First submitted 2020-08-03; First posted 2020-08-25 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Olfaction Disorders; COVID-19
Keywords: anosmia; smell disorder; COVID-19; MRI
MeSH Terms: conditions — Olfaction Disorders; COVID-19; Anosmia | interventions — Olfactometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anosmic or normosmic COVID-19 patients (Other): Patients will undergo ENT exams, olfactometry and MRI.
  Interventions: Diagnostic Test: ENT exam; Diagnostic Test: Olfactometry; Diagnostic Test: Brain MRI

INTERVENTIONS:
Diagnostic Test: ENT exam — ENT examination of the nasal cavity: nasofibroscopy and anterior rhinoscopy.
Diagnostic Test: Olfactometry — Olfactometry test using odorous pens (Sniffin's stick test).
Diagnostic Test: Brain MRI — Brain MRI focused on the olfactory bulbs (3 teslas).

SUMMARY:
Olfactory and gustatory disorders are prevalent symptoms in European COVID-19 patients. This study aimed to detect these disturbances among positive COVID-19 patients (symptom not initially highlighted by the patient and not sought by caregivers) in order to allow early management of olfactory and gustatory dysfunction.

DETAILED DESCRIPTION:
Several medical teams have recently shown that disturbances of smell and taste are common and can be a precursor and even an isolated sign of COVID-19 involvement. Preliminary results suggest the presence of clinical MRI abnormalities, particularly in the olfactory bulbs in anosmic patients with COVID-19.

Anosmia and taste disturbance are early warning signs that could be important in improving the detection and diagnosis of COVID-19, and also in monitoring disease. In addition, disturbances in smell and taste could be an aid in establishing the prognosis of the clinical course of the viral disease. The question of olfactory recovery is also fundamental. To date, we do not know the possibilities of recovery from COVID-19 post viral anosmia. ENT exams, olfactometry and MRI are proposed to study these phenomena.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or over
* Patient with or without a sense of smell diagnosed with a positive COVID-19 PCR test by nasopharyngeal swab in one of the investigation centers
* Patient who has already undergone cerebral MRI and olfactometry, as part of their routine care, within 3 days of being diagnosed with COVID-19+ or who agrees to undergo cerebral MRI and olfactometry within 3 days of being diagnosed with COVID-19+.
* Patient who signed a consent form
* Patient being affiliated to a Health Insurance plan

Exclusion Criteria:

* History of chronic rhino-sinusitis with or without polyp (s)
* History of major craniofacial trauma that led to loss of smell
* History of chronic sense of smell
* Diagnosis of Parkinson's disease or Alzheimer's disease
* Refusal to perform the 3 MRIs
* Refusal to participate in the study
* Pregnant, parturient or lactating woman
* Patient with contraindications to performing MRI
* Patient not speaking or understanding French
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
To compare the qualitative and quantitative morphological abnormalities of the olfactory bulb detected by MRI on initial examination in COVID-19 anosmic versus COVID-19 normosmic patients. | initial examination
  Intensity ratio calculated between average signals of the olfactory bulb and the frontal white matter on a 3-Tesla MRI scanner.
To compare the result of the olfactometry (Sniffin' test) on initial examination in COVID-19 anosmic versus COVID-19 normosmic patients. | initial examination
  Sniffin' test score (T threshold score, D discrimination score, I identification score).

SECONDARY OUTCOMES:
Longitudinal evaluation of qualitative and quantitative abnormalities of olfactory bulbs on MRI in in COVID-19 anosmic patient at initial examination, between 6 weeks and 2 months and between 6 and 9 months. | initial examination, 6 week to 2 months, 6 to 9 months
  Intensity ratio calculated between average signals of the olfactory bulb and the frontal white matter on a 3-Tesla MRI scanner at initial examination, between 6 weeks and 2 months and between 6 and 9 months.
To compare the result of the olfactometry (Sniffin' test) on initial examination in COVID-19 anosmic versus COVID-19 normosmic patients. | initial examination, 6 week to 2 months, 6 to 9 months
  Sniffin' test score (T threshold score, D discrimination score, I identification score).

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Hans, Pr, Study Director — Hopital Foch, Suresnes; Robert-Yves Carlier, Pr, Principal Investigator — Hopital Raymond Poincare, Garches; Jerome Lechien, Dr, Principal Investigator — Hopital Foch, Suresnes
Locations (2):
- France (2):
  - Hopital Raymond Poincare, Garches
  - Hopital Foch, Suresnes, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lechien JR, Chiesa-Estomba CM, De Siati DR, Horoi M, Le Bon SD, Rodriguez A, Dequanter D, Blecic S, El Afia F, Distinguin L, Chekkoury-Idrissi Y, Hans S, Delgado IL, Calvo-Henriquez C, Lavigne P, Falanga C, Barillari MR, Cammaroto G, Khalife M, Leich P, Souchay C, Rossi C, Journe F, Hsieh J, Edjlali M, Carlier R, Ris L, Lovato A, De Filippis C, Coppee F, Fakhry N, Ayad T, Saussez S. Olfactory and gustatory dysfunctions as a clinical presentation of mild-to-moderate forms of the coronavirus disease (COVID-19): a multicenter European study. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2251-2261. doi: 10.1007/s00405-020-05965-1. Epub 2020 Apr 6. PMID 32253535